CLINICAL TRIAL: NCT01297543
Title: A Phase I/II Trial of CLT-008 Myeloid Progenitor Cells in Patients Receiving Chemotherapy for Leukemia or Myelodysplasia
Brief Title: Safety Study of Human Myeloid Progenitor Cells (CLT-008) After Chemotherapy for Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellerant Therapeutics (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CLT008-02
Record Dates: First submitted 2011-02-11; First posted 2011-02-16 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; Myelodysplasia
Keywords: Induction chemotherapy; Re-induction chemotherapy; Consolidation chemotherapy; Leukemia; Myelodysplasia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory, with Excess of Blasts; Leukemia | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Consolidation Group A (Experimental): Low dose CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells; Drug: G-CSF
- Consolidation Group B (Experimental): Intermediate dose CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells; Drug: G-CSF
- Consolidation Group C (Experimental): Intermediate dose CLT-008 (human myeloid progenitor cells), no G-CSF
  Interventions: Biological: human myeloid progenitor cells
- Consolidation Group D (Experimental): High dose CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells; Drug: G-CSF
- Induction Group A1 (cytarabine 7+3) (Active Comparator): G-CSF
  Interventions: Drug: G-CSF
- Induction Group A2 (cytarabine 7+3) (Experimental): Intermediate dose CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells; Drug: G-CSF
- Induction Group A3 (cytarabine 7+3) (Experimental): High dose CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells; Drug: G-CSF
- Induction Group B1 (cytarabine HIDAC) (Active Comparator): G-CSF
  Interventions: Drug: G-CSF
- Induction Group B2 (cytarabine HIDAC) (Experimental): Intermediate dose CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells; Drug: G-CSF
- Induction Group B3 (cytarabine HIDAC) (Experimental): High dose CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells; Drug: G-CSF

INTERVENTIONS:
Biological: human myeloid progenitor cells — Single intravenous injection/infusion
  Other Names: CLT-008; hMPC
  Arms: Consolidation Group A; Consolidation Group B; Consolidation Group C; Consolidation Group D; Induction Group A2 (cytarabine 7+3); Induction Group A3 (cytarabine 7+3); Induction Group B2 (cytarabine HIDAC); Induction Group B3 (cytarabine HIDAC)
Drug: G-CSF — Background therapy
  Other Names: filgrastim; granulocyte colony stimulating factor
  Arms: Consolidation Group A; Consolidation Group B; Consolidation Group D; Induction Group A1 (cytarabine 7+3); Induction Group A2 (cytarabine 7+3); Induction Group A3 (cytarabine 7+3); Induction Group B1 (cytarabine HIDAC); Induction Group B2 (cytarabine HIDAC); Induction Group B3 (cytarabine HIDAC)

SUMMARY:
Ex vivo expanded human myeloid progenitor cells (hMPCs; CLT-008) have the potential to accelerate neutrophil recovery and decrease the risk of febrile neutropenia and infection in patients receiving chemotherapy for acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML), chronic myeloid leukemia (CML), or high-risk myelodysplasia (MDS). In this study, the safety, tolerability and activity of CLT-008 administered after "standard of care" cytarabine-based consolidation or induction/re-induction chemotherapy will be determined by monitoring for adverse reactions, infusion reactions, graft-versus host disease (GVHD), neutrophil and platelet recovery, hMPC persistence, infections and complications.

ELIGIBILITY:
Key Inclusion Criteria:

* Hematological malignancy, including:

  * AML, ALL or MDS
* Planned treatment with cytarabine-based chemotherapy regimen
* Adequate hepatic, renal, hematologic, cardiac and respiratory function

Key Exclusion Criteria:

* Prior allograft or history of active GVHD within 3 years
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse reactions | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose

SECONDARY OUTCOMES:
Duration of neutropenia | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Duration of thrombocytopenia | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Duration of presence of CLT-008 derived cells in blood | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Duration of presence of CLT-008 derived cells in bone marrow | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Incidence of mucositis | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Incidence of infections | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Duration of fever | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Duration of antibiotic use | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Incidence of hospitalization | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose
Duration of hospitalization | Consolidation patients-43 days post dose and Induction/re-induction patients-40 days post dose

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Moores UCSD Cancer Center, La Jolla, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - Loyola University Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplantation, LLC, Beech Grove, Indiana
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Cellerant Therapeutics, Inc. — http://www.cellerant.com